CLINICAL TRIAL: NCT03568786
Title: Influence of the End-inspiratory Pause on Mechanical Ventilation and Its Correlation With Electrical Impedance Tomography
Brief Title: Influence of the End-inspiratory Pause on Mechanical Ventilation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1172-M1-16
Record Dates: First submitted 2018-05-03; First posted 2018-06-26 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Anesthesia; Surgery
Keywords: end-inspiratory pause; lung protection; intraoperative ventilation; lung compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- End-inspiratory pause (EIP) 10% (Experimental): Once the patient is intubated and after initiating ventilation in a volume control mode using a tidal volume of 7 ml/kg of predicted body weight (PBW) with an inspiration: expiration ratio of 1:2; a respiratory rate of 12-14 breaths per minute to maintain the etCO2 at 35-40 mmHg and an initial PEEP of 5 cmH2O, the investigators will apply an alveolar recruitment maneuver (ARM) with estimation of the open lung PEEP using an end-inspiratory pause (EIP) corresponding with a of 10% of the total inspiratory time. Volume control ventilation will be restored after ARM maintaining the same ventilatory parameters except the EIP, which in this group will be of 10% of total inspiratory time.
  Interventions: Procedure: End-inspiratory pause 10%
- End-inspiratory pause (EIP) 30% (Experimental): Once the patient is intubated and after initiating ventilation in a volume control mode using a tidal volume of 7 ml/kg of predicted body weight (PBW) with an inspiration: expiration ratio of 1:2; a respiratory rate of 12-14 breaths per minute to maintain the etCO2 at 35-40 mmHg and an initial PEEP of 5 cmH2O, the investigators will apply an alveolar recruitment maneuver (ARM) with estimation of the open lung PEEP using an end-inspiratory pause (EIP) corresponding with a 30 % of the total inspiratory time. Volume control ventilation will be restored after ARM maintaining the same ventilatory parameters except the EIP, which in this group will be of 30 % of total inspiratory time.
  Interventions: Procedure: End-inspiratory pause 30%

INTERVENTIONS:
Procedure: End-inspiratory pause 10% — Percentage of the total inspiratory time in which there is no gas flow. It is the period of time between the cessation of the inspiratory flow and the start of expiration. In this intervention arm it would correspond to a 10% of the total inspiratory time
  Other Names: Time of inspiratory pause 10%
  Arms: End-inspiratory pause (EIP) 10%
Procedure: End-inspiratory pause 30% — Percentage of the total inspiratory time in which there is no gas flow. It is the period of time between the cessation of the inspiratory flow and the start of expiration. In this intervention arm it would correspond to a 30% of the total inspiratory time
  Other Names: Time of inspiratory pause 30%
  Arms: End-inspiratory pause (EIP) 30%

SUMMARY:
This study evaluates the influence of two different end-inspiratory pause (EIP) times on respiratory mechanics and arterial gases of surgical patients when ventilated under an open lung approach (OLA) strategy. The investigators evaluate the impact of using EIP 10% versus 30% of the inspiratory time on a volume control model. The investigators also analyse the potential influence of these EIP on pulmonary gas distribution measured by electric impedance tomography.

DETAILED DESCRIPTION:
Prolonging the EIP while maintaining an adequate expiratory time has shown benefits in terms of improving alveolar effective ventilation and enhancing gas exchange in surgical and intensive care patients. However, there are no published studies addressing the effects of different EIP times on the respiratory mechanics and gas distribution of surgical patients when associated with OLA strategies for ventilation.

Assuming the benefits of OLA, these investigators hypothesized about the potential effects of increasing the EIP when ventilating patients in a volume control mode. In the present study the investigators evaluated the influence of two different EIP (10% and 30% of the inspiratory time) on the respiratory mechanics of patients submitted to scheduled abdominal surgery under general anesthesia and ventilated with a protective lung strategy. The investigators studied the influence of EIP on driving pressure (Pdriv), plateau pressure (Pplat), respiratory static compliance (Crs) and open lung PEEP (OL-PEEP). We also assessed gas distribution by means of electric impedance tomography and studied its influence on gas exchange measured by means of serial gasometries.

Study protocol. A forced spirometry was performed in all patients after accepting their inclusion.

On the day of surgery, standard monitoring was initiated on arrival in the theatre, including electrocardiography, pulse oximetry, and noninvasive blood pressure monitoring. After light sedation with 1-2 mg of midazolam, a thoracic epidural catheter was placed under local anesthesia on anesthesiologist's criteria. A remifentanil infusion 0.03 mcg/kg/min was started before left radial artery catheterization under local anesthesia. After recording basal data during full consciousness on 21% inspired oxygen, all participants were preoxygenated via a facial mask for 5 min on spontaneous ventilation with fraction of inspired oxygen (FiO2) of 0.7 and fresh gas flow of 6 L/min. After induction with propofol ((1-1.5 mg/kg of predicted body weight (PBW)), 0.8 mg/kg of PBW of rocuronium were administered and proceeded with tracheal intubation. Patients were ventilated via a Primus (Drager, Telford, PA, USA) using a tidal volume of 7 ml/kg of PBW; volume control mode comprised an inspiration: expiration ratio of 1:2 and a respiratory rate of 12-14 breaths per minute to maintain the etCO2 at 35-40 mmHg, with an initial PEEP of 5 cmH2O. EIP was programmed according to randomization group. Fresh gas flow of 2 L/min with FiO2 of 0.7 was used throughout the procedure. Anesthesia was maintained with remifentanil 0.03-0.1 mcg/kg/min and sevoflurane, with minimal alveolar concentration (MAC) of 0.7-1 adjusted for patient´s age. Bispectral Index monitoring was used throughout the entire procedure (BIS Quatro, Covidien Ilc, Mansfield, MA, USA). All ventilation parameters remained stable throughout the study except the EIP (diverted in function of study protocol assignation) and the PEEP, which was tailored according the principles of OLA ventilation previously published. A central venous line was inserted in all cases and continuous cardiac output monitoring, systemic vascular resistance and systolic volume variation were monitored throught out all procedure by means of FloTrac sensor (Edwards Lifesciences, Irvine, California, USA). Other monitoring included train of four (TOF) for neuromuscular relaxation.

Dräger Primus (Dräger Medical, Lübeck, Germany) was used for ventilation with continuous monitoring of peak pressure (Ppk), Pplat, PEEP, Crs, FiO2, fraction of expired oxygen (FeO2), end-tidal CO2 (etCO2). For blood gases an ABL90 FLEX PLUS analyzer (Radiometer Medical, Copenhagen, Denmark) was used. If hemodynamic instability occurred during the ARM (fall> 20% of the cardiac index or mean arterial pressure), maneuver was discontinued and ephedrine or phenylephrine was administered and registered, restoring ARM on haemodynamics recovering.

Ventilatory management Data collection was made in five different moments (moment 0 to 4); moment 0: after endotracheal intubation, on establishing mechanical ventilation and prior to ARM, with the EIP assigned to each group and a standard PEEP of 5 cm H2O. Subsequently an ARM was performed as previously described by Ferrando et al, with calculation of the optimal PEEP by means of a decremental titration trial followed of a new AMR and establishment of a tailored OL-PEEP, 2 cmH2O over optimal PEEP (moment 1). EIP was then crossed between groups (30% in Group 1 and 10% in Group 2), moment 2. Another ARM was then performed with the consequent re-assignation of a different OL-PEEP for each group (moment 3). Finally, EIP was crossed again (moment 4). All data were collected 5 minutes after changes implementation.

Statistic analysis The investigators used the statistical software IBM SPSS Statistics for Windows, version 24 (IBM Corp., Armonk, N.Y., USA) for data analysis. An exploratory analysis of the data was performed using the mean and standard deviation or the median with interquartile ranges for quantitative variables. The investigators used the percentages for analysis of the qualitative variables. The investigators checked the normality of the distribution of data with the Kolmogorov-Smirnov test, or with the Shaphiro-Wilk test for variables with less than 50 records. The Student´s T test for paired samples was used to analyse the difference in the means of quantitative paired variables (intra-group differences), and the Student T test for independent samples to analyse the difference in the means of quantitative variables between both groups (inter-group differences).

Finally, the investigators grouped records corresponding to the EIP applied after recruitment, independently of the original assignation according to Group, In this sense, investigators grouped data corresponding to Group 1 in moment 1 with Group 2 in moment 3 (EIP10% after recruitment) and data of Group 1 in moment 3 with Group 2 in moment 1 (EIP 30% after recruitment), obtaining a sample of 32 registers in comparable paired conditions.

Calculation of the sample size Given the absence of previously published works with an approach similar to the one proposed by investigators, the sample size was calculated based on the data obtained in a pilot sample of 5 patients submitted to surgical and anesthesia management similar to those of the protocol proposed. The investigators estimated the sample size assuming the differences in Crs when changing from an EIP 10 % to 30% in a sequential way (paired sample), determining an average difference 12 ml/cm H2O between both interventions. Sample size was calculated to obtain a power of 80 % to detect differences in the contrast of the null hypothesis h₀: μ₁ = μ₂ by means of a bilateral Student's T test for two related samples, taking into account a level of significance is of 5 %, and assuming a mean of the differences of 12 ± 20 units. Taking into account that the expected percentage of dropouts was 20.00% it would be necessary to recruit 30 pairs of experimental units in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years proposed for major abdominal surgery under general anesthesia.
* Written informed consent.

Exclusion Criteria:

* Participation in another interventional study
* American Society of Anesthesiologists (ASA) classification grade = IV
* Patient in dialysis
* Chronic obstructive pulmonary disease (COPD) grade GOLD (Global Initiative for Chronic Obstructive Lung Disease) > 2
* Functional vital capacity < 60% or > 120% of the predicted
* Body mass index (BMI) > 35 kg/m2
* Relation PaO2/FiO2 <200 mmHg in the baseline sample
* Presence of mechanical ventilation in the 72 hours prior to enrollment
* New York Heart Association (NYHA) functional class ≥ 3
* Clinically suspected heart failure
* Cardiac Index (IC) < 2.5 ml/min/m2 and/or inotropics prior to surgery
* Diagnosis or suspicion of intracranial hypertension
* Presence of pneumothorax or giant bullae on preoperative imaging tests
* Use of Continuous Positive Airway Pressure (CPAP).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Changes in Respiratory System Compliance (ml/cmH2O) | Moment 0 (M0): 5 minutes (min) after tracheal intubation, with volume control and PEEP of 5 cmH2O; M1: 5 min after alveolar recruitment maneuver (ARM); M2: 5 min after crossing time of EIP; M3: 5 min after new ARM; M4: 5 min after crossing time EIP
  Measurement of the respiratory system compliance (Crs; ml/cmH2O) when using an EIP of 10% versus 30% of the global inspiratory time.

SECONDARY OUTCOMES:
Changes in Driving Pressure (Pdriv; cmH2O) | Moment 0 (M0): 5 minutes (min) after tracheal intubation, with volume control and PEEP of 5 cmH2O; M1: 5 min after alveolar recruitment maneuver (ARM); M2: 5 min after crossing time of EIP; M3: 5 min after new ARM; M4: 5 min after crossing time EIP
  Measurement of the Pdriv (cmH2O) when using an EIP of 10% versus 30% of the global inspiratory time.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel López-Herrera, Principal Investigator — Fundación Pública Andaluza para la Investigación de Salud en Sevilla (FISEVI)
Locations (1):
- Fundación Pública Andaluza para la Gestión de Investigación de Salud en Sevilla, Seville, Spain

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
  Study Protocol, Statistical Analysis Plan, Informed Consent Form, Clinical Study Report and Analytic Code will also be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication.and with no end date.
Access Criteria: Researchers who provide a methodologically sound proposal To achieve aims in the approved proposal.
  Proposals should be directed to Dr Daniel López-Herrera; e mail address: dalohero@gmail.com.
  To gain access, data requestors will need to sign a data Access agreement.

REFERENCES:
- [Background] Serpa Neto A, Cardoso SO, Manetta JA, Pereira VG, Esposito DC, Pasqualucci Mde O, Damasceno MC, Schultz MJ. Association between use of lung-protective ventilation with lower tidal volumes and clinical outcomes among patients without acute respiratory distress syndrome: a meta-analysis. JAMA. 2012 Oct 24;308(16):1651-9. doi: 10.1001/jama.2012.13730. PMID 23093163
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Guay J, Ochroch EA. Intraoperative use of low volume ventilation to decrease postoperative mortality, mechanical ventilation, lengths of stay and lung injury in patients without acute lung injury. Cochrane Database Syst Rev. 2015 Dec 7;(12):CD011151. doi: 10.1002/14651858.CD011151.pub2. PMID 26641378
- [Background] Neto AS, Hemmes SN, Barbas CS, Beiderlinden M, Fernandez-Bustamante A, Futier E, Gajic O, El-Tahan MR, Ghamdi AA, Gunay E, Jaber S, Kokulu S, Kozian A, Licker M, Lin WQ, Maslow AD, Memtsoudis SG, Reis Miranda D, Moine P, Ng T, Paparella D, Ranieri VM, Scavonetto F, Schilling T, Selmo G, Severgnini P, Sprung J, Sundar S, Talmor D, Treschan T, Unzueta C, Weingarten TN, Wolthuis EK, Wrigge H, Amato MB, Costa EL, de Abreu MG, Pelosi P, Schultz MJ; PROVE Network Investigators. Association between driving pressure and development of postoperative pulmonary complications in patients undergoing mechanical ventilation for general anaesthesia: a meta-analysis of individual patient data. Lancet Respir Med. 2016 Apr;4(4):272-80. doi: 10.1016/S2213-2600(16)00057-6. Epub 2016 Mar 4. PMID 26947624
- [Background] Amato MB, Meade MO, Slutsky AS, Brochard L, Costa EL, Schoenfeld DA, Stewart TE, Briel M, Talmor D, Mercat A, Richard JC, Carvalho CR, Brower RG. Driving pressure and survival in the acute respiratory distress syndrome. N Engl J Med. 2015 Feb 19;372(8):747-55. doi: 10.1056/NEJMsa1410639. PMID 25693014
- [Background] Ferrando C, Soro M, Canet J, Unzueta MC, Suarez F, Librero J, Peiro S, Llombart A, Delgado C, Leon I, Rovira L, Ramasco F, Granell M, Aldecoa C, Diaz O, Balust J, Garutti I, de la Matta M, Pensado A, Gonzalez R, Duran ME, Gallego L, Del Valle SG, Redondo FJ, Diaz P, Pestana D, Rodriguez A, Aguirre J, Garcia JM, Garcia J, Espinosa E, Charco P, Navarro J, Rodriguez C, Tusman G, Belda FJ; iPROVE investigators (Appendices 1 and 2). Rationale and study design for an individualized perioperative open lung ventilatory strategy (iPROVE): study protocol for a randomized controlled trial. Trials. 2015 Apr 27;16:193. doi: 10.1186/s13063-015-0694-1. PMID 25927183
- [Background] Aguirre-Bermeo H, Moran I, Bottiroli M, Italiano S, Parrilla FJ, Plazolles E, Roche-Campo F, Mancebo J. End-inspiratory pause prolongation in acute respiratory distress syndrome patients: effects on gas exchange and mechanics. Ann Intensive Care. 2016 Dec;6(1):81. doi: 10.1186/s13613-016-0183-z. Epub 2016 Aug 24. PMID 27558174
- [Background] Aboab J, Niklason L, Uttman L, Kouatchet A, Brochard L, Jonson B. CO2 elimination at varying inspiratory pause in acute lung injury. Clin Physiol Funct Imaging. 2007 Jan;27(1):2-6. doi: 10.1111/j.1475-097X.2007.00699.x. PMID 17204030
- [Background] Devaquet J, Jonson B, Niklason L, Si Larbi AG, Uttman L, Aboab J, Brochard L. Effects of inspiratory pause on CO2 elimination and arterial PCO2 in acute lung injury. J Appl Physiol (1985). 2008 Dec;105(6):1944-9. doi: 10.1152/japplphysiol.90682.2008. Epub 2008 Sep 18. PMID 18801962
- [Background] Pillet O, Choukroun ML, Castaing Y. Effects of inspiratory flow rate alterations on gas exchange during mechanical ventilation in normal lungs. Efficiency of end-inspiratory pause. Chest. 1993 Apr;103(4):1161-5. doi: 10.1378/chest.103.4.1161. PMID 8131458
- [Background] Aboab J, Niklason L, Uttman L, Brochard L, Jonson B. Dead space and CO(2) elimination related to pattern of inspiratory gas delivery in ARDS patients. Crit Care. 2012 Dec 12;16(2):R39. doi: 10.1186/cc11232. PMID 22390777
- [Background] Fuleihan SF, Wilson RS, Pontoppidan H. Effect of mechanical ventilation with end-inspiratory pause on blood-gas exchange. Anesth Analg. 1976 Jan-Feb;55(1):122-30. doi: 10.1213/00000539-197601000-00034. PMID 942823
- [Background] Astrom E, Uttman L, Niklason L, Aboab J, Brochard L, Jonson B. Pattern of inspiratory gas delivery affects CO2 elimination in health and after acute lung injury. Intensive Care Med. 2008 Feb;34(2):377-84. doi: 10.1007/s00134-007-0840-7. Epub 2007 Sep 1. PMID 17763841
- [Background] Suter PM, Jevic MG, Hemmer M, Gemperle M. [The effects of the pause at the end of inspiration on gas exchange and hemodynamics during artificial ventilation]. Can Anaesth Soc J. 1977 Sep;24(5):550-8. doi: 10.1007/BF03005528. French. PMID 332285
- [Background] Bardoczky GI, d'Hollander AA, Rocmans P, Estenne M, Yernault JC. Respiratory mechanics and gas exchange during one-lung ventilation for thoracic surgery: the effects of end-inspiratory pause in stable COPD patients. J Cardiothorac Vasc Anesth. 1998 Apr;12(2):137-41. doi: 10.1016/s1053-0770(98)90319-6. PMID 9583541
- [Background] Sturesson LW, Malmkvist G, Allvin S, Collryd M, Bodelsson M, Jonson B. An appropriate inspiratory flow pattern can enhance CO2 exchange, facilitating protective ventilation of healthy lungs. Br J Anaesth. 2016 Aug;117(2):243-9. doi: 10.1093/bja/aew194. PMID 27440637
- [Background] Taskar V, John J, Larsson A, Wetterberg T, Jonson B. Dynamics of carbon dioxide elimination following ventilator resetting. Chest. 1995 Jul;108(1):196-202. doi: 10.1378/chest.108.1.196. PMID 7606958
- [Derived] Lopez-Herrera D, De La Matta M. Influence of the end inspiratory pause on respiratory mechanics and tidal gas distribution of surgical patients ventilated under a tailored open lung approach strategy: A randomised, crossover trial. Anaesth Crit Care Pain Med. 2022 Apr;41(2):101038. doi: 10.1016/j.accpm.2022.101038. Epub 2022 Feb 17. PMID 35183806